CLINICAL TRIAL: NCT04683796
Title: Comparison of Treatment Efficacy Between 100% Platelet-rich Plasma and 100% Serum Eye Drops in Moderate to Severe Dry Eye Disease: A Randomized Controlled Trial Protocol
Brief Title: Comparison of Efficacy Between 100% Platelet-rich Plasma and 100% Serum Eye Drops in Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Passara Jongkhajornpong, Department of Ophthalmology, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1996
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either 100% APRP or 100% AS (the same treatment for both eyes).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment package will be labelled as randomization number. Participants will also be blinded to the treatments they receive by using the identical type of eye drop bottle. Clinical and research staffs involved in the outcome assessments will be blinded to the treatment allocation. Lastly, data analysts will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100% APRP (Experimental): Patients will be instructed to apply every 2 hours (8 times/day). The currently used bottle will be required to store at 4 C for 24 hours, and the remaining bottles at -20 C in a freezer until day of use.
  Interventions: Drug: 100% Autologous platelet rich plasma
- 100% AS (Active Comparator): Patients will be instructed to apply every 2 hours (8 times/day). The currently used bottle will be required to store at 4 C for 24 hours, and the remaining bottles at -20 C in a freezer until day of use.
  Interventions: Drug: 100% Autologous serum

INTERVENTIONS:
Drug: 100% Autologous platelet rich plasma — Patients' blood (36 ml per tube) will be collected in three 50-ml sterile centrifuge tubes containing 4 ml of 3.2% buffered citrate acid for anticoagulation. Tubes will be centrifuged at 350 g for 10 minutes at 20 C. The two upper layers of the centrifuged blood, the plasma and the superficial buffy coat, will be separated in a sterile manner under a laminar air flow hood. A 1.5 ml aliquot of both final blood products will be transferred into identical opaque eye drop bottles, labelled name, hospital number, dated and sealed.
  Other Names: APRP
  Arms: 100% APRP
Drug: 100% Autologous serum — Patients' blood (36 ml per tube) will be collected in three 50-ml sterile centrifuge tubes. The tubes will be left standing in an upright position for 1-2 hours to enable blood clot formation at room temperature (18-25 C). The tubes will be centrifuged at 3000 g for 30 minutes at 20 C. The supernatant serum will be aseptically transferred into a sterile syringe to enable filtration through a 0.2 µm pore size membrane filter under a laminar air flow hood. A 1.5 ml aliquot of both final blood products will be transferred into identical opaque eye drop bottles, labelled name, hospital number, dated and sealed.
  Other Names: AS
  Arms: 100% AS

SUMMARY:
Dry eye disease (DED) is a common eye problem, affecting 5% to 50% of the world population. Although the disease is not fatal, it substantially reduces quality of life and creates a high economic burden as high as over 50 billion from a societal perspective. Several biological tear substitutes (e.g., autologous serum (AS), autologous platelet rich plasma (APRP), and autologous platelet lysate (APL)) could effectively improve dry eyes, especially in patients with moderate to severe DED.. However, evidence on their comparative efficacy is controversial. The objective of the study is to compare the efficacy of 100% APRP with 100% AS eye drops in patients with moderate to severe DED.

DETAILED DESCRIPTION:
The study is a single-center, double-blinded randomized, parallel, non-inferiority trial. Patients will be recruited from out-patient clinic, Department of Ophthalmology, Ramathibodi Hospital, Bangkok and will be randomized to receive either 100% APRP or 100% AS eye drops (1:1 ratio) for 4 weeks. The primary outcomes include ocular surface disease index (OSDI) and ocular surface staining evaluated using the Oxford scale. Secondary outcomes are fluorescein break-up time (FBUT), Schirmer's I test (ST I), meibomian gland parameters and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to less than 75 years.
* Have OSDI scores ≥ 23 or Oxford staining grade ≥ 2.
* Do not have following conditions:

Uncontrolled systemic diseases, active infection, advanced cancer. Pregnant and nursing women. • Have not recently used the following medications/interventions/surgery: Anticoagulants or anti-platelets. Topical undiluted blood products within 3 months. Punctal plug or contact lenses. Ocular surgery within 6 months.

* Do not have active ocular infection/inflammation, abnormal eyelid function or severe meibomian gland dysfunction (MGD stage 4).
* Have no contraindication for blood donations:

Positive human immunodeficiency virus, hepatitis B or C, or syphilis. Anemia (Hb < 11 g/dL) or platelet concentration < 150,000/ml.

* Being able to stop current dry eye treatment for 48 hours before staring trial intervention
* Willing to comply with the 4-week study protocol and provide informed consent.

Exclusion Criteria:

• None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Ocular surface score index (OSDI) | 4 weeks
  The OSDI is a patient-reported outcome (PRO) questionnaire which was designed by Allergan, Inc. to assess range of ocular symptoms related to chronic dry eye disease and reflect patient's ability of function. It comprised 12 questions which are divided into 3 subscales including ocular symptoms (5 questions), vision-related function (4 questions), and environmental triggers (3 questions). Each of question is rated from 0 to 4 indicating none of the time, some of the time, half of the time, most of the time and all of the time, respectively. The average OSDI is transformed into a score ranged from 0 to 100, with a higher score indicating more severity of dry eye disease. The OSDI is classified as normal (0-12 points), mild (13-22 points), moderate (23-32 points) and severe (33-100).
Ocular surface staining (OSS) | 4 weeks
  To assess total ocular surface staining, the cornea and conjunctival staining are graded by using Oxford scale guidelines (range grade 0 to 5). The higher score refers to higher severity of dry eye.

SECONDARY OUTCOMES:
Fluorescein break up time (FBUT) | 4 weeks
  The break up time (seconds) will be measured after fluorescein staining by using a stopwatch starting from the time of complete eye lid opening to the time of the first tear break up appear. The average values of 3 times of FBUT will be used. The reference value for DED diagnosis is used ranged from a cut-off time of less than 10 seconds for dry eye and less than 5 seconds for severe dry eye.
Schirmer's test (ST) | 4 weeks
  The Schirmer test (ST) was performed using commercially available prepackaged sterile paper strips without anesthesia. The rounded bulb end of the strip was folded and placed in the lateral canthus away from the cornea and left in place for 5 minutes after which the wet strip length was recorded in mm. Tear deficiency is defined if ST is less than 5 mm wetting of the paper after 5 minutes.
Meibum quality and expressibility. | 4 weeks
  Meibum quality is assessed by applying the pressure on each of 8 glands of the central third of the lower lid on a scale of 0 to 3 for each gland: 0, clear; 1, cloudy; 2, cloudy with debris (granular); and 3, thick, like toothpaste (total score range, 0-24). Higher score indicates the higher severity of meibomian gland dysfunction.
  Expressibility is assessed on a scale of 0 to 3 in five glands in the lower or upper lid, according to the number of glands expressible: 0, all glands; 1, three to four glands; 2, one to two glands; and 3, no glands. Higher score indicates the higher severity of meibomian gland dysfunction.
Number of patients with ocular adverse events | 4 weeks
  All ocular adverse events will be recorded throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ammarin Thakkinstian, Ph.D., Study Director — Department of Clinical Epidemiology and Biostatistics, Mahidol University, Thailand
Locations (1):
- Ophthalmology Department, Ramathibodi Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Data will be available upon the specific request.

REFERENCES:
- [Derived] Jongkhajornpong P, Lekhanont K, Rattanasiri S, Pisitkun P, Thakkinstian A. Comparison of Corneal Epitheliotrophic Factors of Undiluted Autologous Platelet-Rich Plasma and Autologous Serum Eye Drops for Dry Eye Disease. Ophthalmol Ther. 2025 Feb;14(2):363-377. doi: 10.1007/s40123-024-01082-y. Epub 2024 Dec 20. PMID 39704778
- [Derived] Jongkhajornpong P, Lekhanont K, Rattanasiri S, Numthavaj P, McKay G, Attia J, Thakkinstian A. Efficacy of 100% autologous platelet-rich plasma and 100% autologous serum in dry eye disease: a randomised controlled trial. BMJ Open Ophthalmol. 2024 Oct 8;9(1):e001857. doi: 10.1136/bmjophth-2024-001857. PMID 39384222
- [Derived] Jongkhajornpong P, Numthavaj P, Anothaisintawee T, Lekhanont K, McKay G, Attia J, Thakkinstian A. Comparison of treatment efficacy between 100% platelet-rich plasma and 100% serum eye drops in moderate-to-severe dry eye disease: a randomised controlled trial protocol. BMJ Open. 2021 Jun 30;11(6):e048479. doi: 10.1136/bmjopen-2020-048479. PMID 34193498